CLINICAL TRIAL: NCT04466254
Title: A Phase II Study Evaluating the Efficacy and Safety of Combination of CPGJ602 and Chemotherapy as First Line Treatment in KRAS/NRAS/BRAF Wild-type, Metastatic Colorectal Cancer Patients
Brief Title: Efficacy and Safety Study of Combination of CPGJ602 and Chemotherapy, in First Line, With Wild KRAS/NRAS/BRAF in Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-602-mCRC-II-01
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): CPGJ602 325mg/m2 IV Q2W； mFOLFOX6 therapy starts on day 1 and ends on day 2, then repeats every 2 weeks.
  Interventions: Drug: CPGJ602
- Arm B (Experimental): CPGJ602 400 mg/m2 IV in the first infusion， then 250mg/m2 followed per every week； mFOLFOX6 therapy starts on day 1 and ends on day 2, then repeats every 2 weeks
  Interventions: Drug: CPGJ602
- Arm C (Active Comparator): cetuximab 400 mg/m2 IV in the first infusion， then 250mg/m2 followed per every week； mFOLFOX6 therapy starts on day 1 and ends on day 2, then repeats every 2 weeks
  Interventions: Drug: cetuximab

INTERVENTIONS:
Drug: CPGJ602 — Q2W/QW iv
  Arms: Arm A; Arm B
Drug: cetuximab — QW iv
  Arms: Arm C

SUMMARY:
To assess the efficacy and safety of the combination of CPGJ602 and chemotherapy in subjects with KRAS/NRAS/BRAF wild-type, metastatic colorectal cancer.

DETAILED DESCRIPTION:
This is an open label, randomized, positive control, phase II study to treat subjects with KRAS/NRAS/BRAF wild-type, unresectable metastatic colorectal cancer. The patients will be randomized into three arms consist of CPGJ602 (2 weeks/cycle) + mFOLFOX6, CPGJ602 (1 week/cycle) + mFOLFOX6, and cetuximab (1 week/cycle) + mFOLFOX6 at a ratio of 2:2:1. This study is conduct to assess the efficacy and safety of three treatments for patients.

ELIGIBILITY:
Inclusion Criteria:

* informed consent to study procedures, male or female， 18-80 years old.
* Histologically or cytologically proven diagnosis of unresectable metastatic colorectal cancer
* Patients were confirmed by central lab with KRAS, NRAS and BRAF wild type. All patients must undergo a fresh tumor biopsy during the screening process, or provide archived tumor samples
* EOCG: 0~1 within 7 days prior to first treatment
* Life expectancy of at least 3 months
* Patients must have adequate hematology, liver and kidney function, (had been received no blood transfusion, albumin, recombinant human thrombopoietin or colony stimulating factor therapy, renal replacement therapy, etc. within 14 days prior to the first study drug therapy, and the laboratory tests met the following requirements):

Hepatic: white blood count (WBC)≥ 3.0 × 109, absolute neutrophil count (ANC)≥ 1.5 x 109/L, platelet count (PLT)≥ 100 x 109/L, haemoglobin (Hb) ≥ 90 g/dL.

Liver: total bilirubin (T-Bil)≤ 1.5 times the upper limit of normal (ULN), aspartate transaminase (AST) and/or alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤5 × ULN if with liver involvement) Kidney: Serum albumin ≥28 g/L, urea nitrogen 1.5 ×the ULN (If the center cannot detect BUN, it could be substituted by detecting urea), serum creatinine ≤1.5 × the ULN or creatinine clearance≥50mL/min

* According to RECIST1.1, the subject should have an assessable lesion
* Able to understand and willing to sign the Informed Consent Form (ICF)
* Patients with good compliance assessed by investigator

Exclusion Criteria:

* Those who have received any previous anti-tumor therapy such as salvage chemotherapy, targeted therapy, biological immunotherapy, etc. (The treatment of adjuvant, neoadjuvant and radiotherapy sensitized chemotherapy discontinued 6 months or more [platinum containing chemotherapy should be treated for at least 12 months]. Patients with disease progression can be enrolled and chemotherapy-related toxicity should be restored to grade 1 or below [except for hair loss])
* Patients who have had surgery within 28 days prior to first treatment with the study drug. While, those who had primary excision or palliative ostomy with good recovery within 14 days before receiving the first study drug
* Those who received radiotherapy within 28 days prior to first dose of study drug, while those who received palliative radiotherapy and recovered well within 14 days prior to receiving the study drug
* Patients with other serious uncontrolled disease (e.g. interstitial pneumonia, epilepsy, hepatic failure, etc)
* Patients had other active malignant tumor, except for the followings:

The under-treated non-melanoma skin cancer;Cured cervical cancer or basal cell carcinoma of the skin, mammary gland ductal carcinoma in situ, and phase 1, grade 1 endometrial carcinoma

* Patients infected as followings; Hepatitis B: HBV DNA titer> 2000 IU/ml; Hepatitis C: HCV RNA titer>ULN; HIV infection; Serious bacterial infection; Active mycobacterium tuberculosis infection; Serious other active microbial and parasitic infections.
* History of psychiatric, psychological illness (except for those patients whose mild mental illness have been cured for more than 3 years and have no signs of recurrence assessed by the researchers), or had history of alcohol or drug abuse
* Known or suspected to have brain metastases and/or cerebrospinal meningitis
* Patients with acute or subacute intestinal obstruction, or with a history of inflammatory bowel disease， or who had gastrointestinal perforation and unhealed
* Patients with serious cardiovascular and cerebrovascular diseases，these include but are not limited to the followings:

Patients with uncontrolled hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg under regular drug control); Patients with hypertensive crisis or had a history of hypertensive encephalopathy; Cerebrovascular accidents, transient ischemic attacks and myocardial infarction within 6 months prior to treatment with the study drug, and significant vascular disease (including, but not limited to, aortic aneurysms or proximal arterial thrombosis requiring surgical repair); Unstable angina; Heart failure (NYHA ≥Ⅱ) Uncontrolled serious arrhythmia by drug (ECG QTc ≥450ms for male, and QTc≥470ms for female, calculated by Fridericia formula)

* Patients with thrombotic dysfunction: International standardized ratio (INR) or activated partial thromboplastin time APTT, any of which ≥1.5×ULN
* Patients who are known to be allergic to the study drug or its excipients, or have a history of severe allergies to other monoclonal antibodies
* Patients who are in pregnant or breastfeeding, or are unable to use reliable contraception during the study and 6 months after discontinued treatmen
* Patients received any experimental drug in other interventional clinical trials: the time from stopping taking the study drug of a previous treatment to take the first dose of this study drug is less than 28 days or less than 5 half-lives of the drug, whichever is longer
* Patients who have a history of organ transplant, including autologous/allogeneic stem cell transplantation
* Patients who have a history of severe dry eye and Patients who Currently suffering from severe dry eye disease , keratitis,and ulcerative keratitis.
* Other conditions which are not fit for this study assessed by investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Best of Response (BOR) | for 16 weeks
  Defined as the percentage of patients whose overall response is CR or PR from day 1 to 16th week of study and maintain at least until efficacy confirmation assessment (4 weeks ± 2 days), per RECIST v1.1 for target lesions assessed by BIRC.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | for 16 weeks
  Defined as the interval from the date of randomization until first documented disease progression or death from any cause, whichever occurs first, assessed based on tumor assessments according to RECIST v1.1 per BICR and Investigator.
BOR Assessed by investigator | for 16 weeks
Disease Control Rate (DCR) | for 16 weeks
  Defined as the percentage of patients whose overall response is CR, PR and SD from day 1 to 16th week and maintain at least until efficacy confirmation assessment (4 weeks ± 2 days), per RECIST v1.1 for target lesions assessed by BIRC and Investigator.
unConfirmed BOR at the end of 16th week by BICR and Investigator. | for 16 weeks
  Defined as the percentage of patients whose overall response is CR or PR from day 1 to 16th week per RECIST v1.1 for target lesions assessed by BIRC and Investigator.
Time to Tumor Response (TTR) | for 16 weeks
  Defined as the time from the first dose study treatment until the date of the first assessment of confirmed CR or PR, assessed by BICR and Investigator
Deepness of Response (DpR) | for 16 weeks
  The relative change in the sum of longest diameters of RECIST target lesions at the nadir, in the absence of new lesions or progression of non-target lesions, when compared with baseline assessed by BIRC and Investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China